CLINICAL TRIAL: NCT03662932
Title: Early Intensive Mobilization Following Acute High-risk Abdominal Surgery - a Feasibility Study
Brief Title: Early Mobilization Following Emergency Abdominal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Morten Tange Kristensen PT, PhD (Other)
Responsible Party: Sponsor-Investigator, Morten Tange Kristensen PT, PhD, Senior researcher, PT, Phd, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HH-AHA-FYS-02
Record Dates: First submitted 2018-08-23; First posted 2018-09-10 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Acute High-risk Abdominal Surgery (AHA)
Keywords: Abdominal surgery; Early mobilization; Feasibility

STUDY DESIGN:
Intervention Model Description: All the included participants receive the intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early intensive mobilization (Experimental): Progressed mobilization from postoperative day 0.
  Interventions: Other: Early intensive mobilization

INTERVENTIONS:
Other: Early intensive mobilization — Early mobilization: mobilization with the hospital staff begins already on the day of surgery, and includes mobilization in and out of bed, rise up from a chair, standing and walking.
  Intensive mobilization: mobilization more than 4 times a day in the first postoperative week.

SUMMARY:
Acute High-risk abdominal surgery (AHA) is associated with high mortality rates, multiple postoperative complications and prolonged duration of hospital admission. A recent study revealed very low level of physical performance in the first postoperative week in patients undergoing AHA. Furthermore the included patients who were non-independently mobilized or had low level of 24-hour physical activity more often experienced a pulmonary complication. Studies examining the feasibility of early and intensive mobilization are needed, prior to investigating the effect of the intervention in an Randomised Controlled Trial. The purpose of this study is evaluating the feasibility of early and intensive mobilization during the first week postoperatively among patients who receive Acute High-Risk Abdominal Surgery (AHA). The aim is also to describe physical performance, physical activity, pulmonary function and health-related quality of life, as well as barriers to mobilization following AHA surgery.

ELIGIBILITY:
Inclusion Criteria:

• Patients (18 years and older) undergoing emergency laparotomy or laparoscopy (inclusive reoperations after elective surgery).

Exclusion Criteria:

* Patients undergoing minor emergency operations (uncomplicated appendectomy, laparoscopic cholecystectomy, diagnostic laparoscopy or laparotomy without intervention).
* Patients not able to give consent to participation in the study within 48 hours after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2018-12-21 (Actual)

PRIMARY OUTCOMES:
Mobilization within 24 hours after surgery assessed by CAS | Up to 24 hours after surgery
  Percentage of participants that is mobilized within 24 hours after surgery assessed by the Cumulated Ambulation Score (CAS).
  Pre-defined criteria of feasibility; >=80% feasible, 60-79% potentially feasible, and <60% considered not feasible.
Time out of bed (minutes per day) assessed by a accelerometer | Up to 7 days after surgery
  Percentage of participants able to meet the predefined daily targets of time out of bed (minutes per day) assessed by a accelerometer recording time spent in lying, sitting and standing/walking.
  Pre-defined criteria of feasibility; >=80% feasible, 60-79% potentially feasible, and <60% considered not feasible.
Mobilization 4 times a day registered in a journal | Up to 7 days after surgery
  Percentage of participants mobilized 4 times a day registered by the hospital staff in a journal.
  Pre-defined criteria of feasibility; >=80% feasible, 60-79% potentially feasible, and <60% considered not feasible.
Able to complete the outcome measures: NRS, VAFS, CST, Peakflow and EQ-5D-5L | Up to 7 days after surgery
  Percentage of participants able to complete the selected outcome measures: Numeric Rating scale (NRS), Visual Analog Fatigue Scale (VAFS), 30-second Chair Stand Test (CST), Peakflow meter and health-related quality of life EQ-5D-5L.
  Pre-defined criteria of feasibility; >=80% feasible, 60-79% potentially feasible, and <60% considered not feasible.

SECONDARY OUTCOMES:
Postoperative Pulmonary complication | Up to 2 weeks after surgery
  The occurrence of postoperative pulmonary complication defined as Clavien-Dindo classification higher than grade 1
Cumulated Ambulation Score (CAS, 0-6 points) | Up to 7 days after surgery
  Evaluation of independence in basic mobility (in and out of bed, rise from a chair and walking). Scale range is 0-6 points: 0 points indicate that the participant can't be mobilized and 6 points indicate that the participant is mobilizied independently.
Functional independence in Activity of Daily Living assessed by Barthel Index (BI, 0-100 points) | Up to 7 days after surgery
  Measure functional independence in Activity of Daily Living (ADL) in relation to transfer, mobility, stairs, dressing, feeding, grooming, bathing, toilet use and bowels and bladder function. Scale range is 0-100 points and lower scores indicates increased disability.
30-second Chair Stand Test (CST) | Up to 7 days after surgery
  Test for lower body leg strength and endurance assessed by the 30-second Chair Stand Test (CST). Record the number of times the patient stands in 30 sec.
24-hour physical activity (minutes per day) | Up to 7 days after surgery
  Accelerometer recording time spent in lying, sitting and standing/walking.
Pulmonary function assessed by Peak flow meter | Up to 7 days after surgery
  Measure of a participants maksimum speed of exspiration assessed by a peak flow meter
Visual Analog Fatigue Scale (VAFS, 0-10 points) | Up to 7 days after surgery
  Intensity of fatigue after surgery. Scale range is 0-10 points and higher scores indicate higher degree of fatigue.
Pain assessed by Numeric Rating scale (NRS, 0-10 points) | Up to 7 days after surgery
  Self-reported measure of pain intensity. Scale range is 0-10 points and higher scores indicate higher degree of pain.
Health-related quality of life assessed by EQ-5D-5L (0-100 points) | Up to 7 days after surgery
  Standardized instrument developed by the EuroQol Group as a measure of self-reported health-related quality of life. Scale range is 0-100 points: 0 points indicating the worst health the participant can imagine.

OTHER OUTCOMES:
Barriers to mobilization | Up to 7 days after surgery
  Self-reported barriers to mobilization during hospitalization.
Pre-hospital functional level assessed by New Mobility Score (NMS, 0-9 points) | Baseline
  Measure of pre-hospital walking functional level. Scale range is 0-9 points: higher scores indicating independent level of walking ability.

CONTACTS AND LOCATIONS:
Overall Officials: Morten T Kristensen, PhD, Study Chair — Hvidovre University Hospital
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark